CLINICAL TRIAL: NCT01512693
Title: Single Dose Study to Investigate the Pharmacokinetics of Odanacatib (MK-0822) in Subjects With Hepatic Insufficiency
Brief Title: Assessment of Pharmacokinetics of Single Dose Odanacatib (MK-0822) in Participants With Moderate Hepatic Insufficiency (MK-0822-070)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0822-070
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — odanacatib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Hepatic Insufficiency Group (Experimental): Single-dose administration of odanacatib 50 mg to participants with moderate hepatic insufficiency.
  Interventions: Drug: MK-0822
- Healthy Matched Control Group (Experimental): Single-dose administration of odanacatib 50 mg to healthy matched control participants.
  Interventions: Drug: MK-0822

INTERVENTIONS:
Drug: MK-0822 — A single oral dose (50 mg tablet) of MK 0822 will be administered on Day 1 after an overnight fast.
  Other Names: odanacatib

SUMMARY:
This open-label, non-randomized study was designed to compare pharmacokinetics of a single 50 milligram (mg) dose of MK-0822 in participants with and without moderate hepatic insufficiency (abnormal liver function) in order to determine to what degree hepatic dysfunction may impact therapeutic blood levels of MK-0822. The primary hypothesis is that plasma AUC0-∞ of odanacatib in participants with moderate hepatic insufficiency is similar to that in matched healthy participants following a single 50 mg oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Not currently pregnant, nursing or planning to be pregnant through-out the course of the study; agree to use specified contraception per protocol requirement
* Body Mass Index (BMI) of ≤ 39 kg/m^2 (not obese)
* Judged to be in good health (for healthy participant population)
* Non-smoker for the past 6-months; social smokers (smoke less than 10 cigarettes within the past 3 months; or per discretion of the study Investigator, quit smoking within the past 3 months.
* Diagnosed with chronic (more than 6 months), stable (no acute episodes of illness within the previous 2 months) hepatic insufficiency (liver dysfunction) with features of cirrhosis due to any cause (for the moderate hepatic insufficiency participant population)
* Possess the ability to understand the study, grant voluntary informed consent and willingly comply with all study requirements

Exclusion Criteria:

* Does not meet the age requirement, is mentally or legally incapacitated, has or is expected to have significant emotional problems, or a history of a clinically significant psychiatric disorder
* Has been diagnosed with a disease or medical condition which may pose a risk to the participant or may confound the study results
* Compromised renal (kidney) function, significant organ system disease(s) or cancer(s)
* Unable to refrain from or anticipates the use of any new medication, including prescription and non-prescription drugs or herbal remedies
* Meets the requirements of the study in regard to current medication profile including: prescribed medications, caffeine, alcohol, over-the-counter drugs, herbals and nutritional products; with expected non-use of recreational (illicit) drugs associated with misuse, abuse and/or addiction
* Had surgery, donated 1 unit of blood or received another investigational study medication within 4 weeks prior to the study's first dose of investigational product
* History of multiple and/or severe allergies, or has had a life-threatening reaction or inability to tolerate prescription or non-prescription drugs or food

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-02-23 (Actual); Primary Completion 2012-04-24 (Actual); Study Completion 2012-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Hepatic Insufficiency Group | Healthy Matched Control Group
Started | 8 | 9
Completed | 8 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Insufficiency Group | Healthy Matched Control Group | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (4.9) | 54.2 (5.3) | 53.7 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of MK-0822 From Time 0 to Infinity (AUC0-∞) After Single Dose
Description: For healthy and moderate hepatic insufficiency participants, plasma samples were collected from predose to 336 hours postdose for determination of AUC0-∞ (Total AUC). AUC0-∞ is a measure of total drug exposure.
Time Frame: Pre-dose and 1, 2, 4, 6, 9, 12, 16, 24, 32, 48, 72, 96, 120, 168, 240, and 336 hours postdose
Population: The per protocol population consisted of all participants who complied with the protocol sufficiently to ensure that results will likely exhibit the effects of treatment according to the underlying scientific model.
Measure: Least Squares Mean (95% Confidence Interval); unit: μM*hr
Arm/Group | Moderate Hepatic Insufficiency Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
μM*hr | 28.84 [21.88 to 38.01] | 33.79 [25.64 to 44.54]
Statistical Analysis 1: Comparison: Moderate Hepatic Insufficiency Group vs Healthy Matched Control Group; Natural log-transformed plasma values were analyzed using an analysis of covariance (ANCOVA) model with a categorical factor for population (moderate hepatic insufficiency participants, healthy matched control participants) and continuous covariates for age and body mass index (BMI). Data are back transformed to geometric least-squares mean ratio (GMR) (moderate hepatic insufficiency / healthy) and 90% confidence intervals; Test type: Non-Inferiority or Equivalence — Similarity will be concluded if the GMR (moderate hepatic insufficiency / healthy) is contained within the interval [0.40, 2.50]; GMR = 0.85, 90% CI 2-sided [0.61 to 1.19]

2. Secondary Outcome: Maximum Concentration (Cmax) of MK-0822 After Single Dose
Description: For healthy and moderate hepatic insufficiency participants, plasma samples were collected from predose to 336 hours postdose for determination of Cmax.
Time Frame: Pre-dose and 1, 2, 4, 6, 9, 12, 16, 24, 32, 48, 72, 96, 120, 168, 240, and 336 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate Hepatic Insufficiency Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
nM | 199.41 [150.26 to 264.64] | 279.59 [210.68 to 371.05]
Statistical Analysis 1: Comparison: Moderate Hepatic Insufficiency Group vs Healthy Matched Control Group; Natural log-transformed plasma values were analyzed using an ANCOVA model with a categorical factor for population (moderate hepatic insufficiency participants, healthy matched control participants) and continuous covariates for age and BMI. Data are back transformed to GMR (moderate hepatic insufficiency / healthy) and 90% confidence intervals; Test type: Superiority or Other; GMR = 0.71, 90% CI 2-sided [0.51 to 1.00]

3. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-0822 After Single Dose
Description: For healthy and moderate hepatic insufficiency participants, plasma samples were collected from predose to 336 hours postdose for determination of Tmax.
Time Frame: Pre-dose and 1, 2, 4, 6, 9, 12, 16, 24, 32, 48, 72, 96, 120, 168, 240, and 336 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Moderate Hepatic Insufficiency Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
hr | 4.00 [2.00 to 48.00] | 24.00 [2.00 to 48.00]

4. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MK-0822 After Single Dose
Description: Apparent terminal half-life is the time required to divide the plasma (serum) concentration by two after reaching pseudo-equilibrium. (Note: it is not the time required to eliminate half the administered dose.) For healthy and moderate hepatic insufficiency participants, plasma samples were collected from predose to 336 hours postdose for determination of t1/2. Results are presented using harmonic mean and jackknife standard deviation.
Time Frame: Pre-dose and 1, 2, 4, 6, 9, 12, 16, 24, 32, 48, 72, 96, 120, 168, 240, and 336 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Moderate Hepatic Insufficiency Group | Healthy Matched Control Group
Number analyzed (Participants) | 8 | 8
hr | 91.5 (30.1) | 70.5 (10.2)

ADVERSE EVENTS:
Time Frame: Up to 15 days
Description: The safety population consisted of all participants who received at least one dose of the study drug.
Arm/Group | Moderate Hepatic Insufficiency Group | Healthy Matched Control Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 1/8 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Insufficiency Group (N=8) | Healthy Matched Control Group (N=9)
Nasopharynigitis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days